CLINICAL TRIAL: NCT04936737
Title: The Influence of Exercise on Tissue Beta-alanine Uptake and Carnosine Synthesis Rates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Gualano, Professor, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B-alanine and HIIT
Record Dates: First submitted 2021-04-16; First posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Exercise Training; Carnosine; Dietary Supplements
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: The order of treatments will be random
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beta-alanine supplementation and high intensity exercise (Experimental): Individuals will participate in a high-intensity exercise and will be supplemented with beta-alanine. This protocol will be conducted for six non-consecutive days.
  Interventions: Dietary Supplement: Beta-alanine supplementation; Other: High intensity interval exercise
- Beta-alanine supplementation only (Experimental): In this protocol, the individuals will be supplemented with beta-alanine without the exercise protocol for six non-consecutive days.
  Interventions: Dietary Supplement: Beta-alanine supplementation

INTERVENTIONS:
Dietary Supplement: Beta-alanine supplementation — The supplementation will be administrated in the dosage of 20mg.kg-1. On the first and the sixth (last one), one dose of beta-alanine will be taken. On the other four days of supplementation, the volunteers will take 2 doses (20mg.kg-1) of Beta-alanine.
Other: High intensity interval exercise — The HIIE sessions will consist of 10 series of 1 min of effort, divided into two blocks of 5 series each. There will be an interval of 5 min of passive recovery; within each block, the interval between sets will be 1 min of active recovery. The exercise will be conducted in a mechanical brake cycle ergometer, with load applied by placing washers on a load plate (Biotec 2100, Cefise, Brazil).
  Arms: Beta-alanine supplementation and high intensity exercise

SUMMARY:
B-alanine supplementation is highly efficient in increasing intramuscular carnosine content, leading to improved physical performance, especially in high-intensity exercises (HIIE). It seems that exercise per se can modulate carnosine content; however, it remains uncertain whether physical training or training status can influence B-alanine supplementation responses. Thus, this work aims to assess whether HIIE can increase B-alanine uptake by peripheral tissues and, more specifically, skeletal muscle and increase intramuscular carnosine synthesis. The volunteers will be evaluated in two conditions: intake of B-alanine + exercise (B-EX) and B-alanine intake only (B-Ala). This process will be divided into two blocks of six days (Thursday to Thursday - without the weekend) with a 4-6 weeks washout. In the B-EX block, a 20-minute HIIE session will be held. In the B-Ala block, the same procedures will be adopted for the B-EX block, with the replacement of the HIIE for 20 minutes of rest sitting on the cycle ergometer. We will evaluate the determination of muscle B-alanine, plasma, and urine, the gene expression of carnosine-related enzymes and transporters, the enzymes Carnosine Synthase 1 (CARNS1), carnosine dipeptidase 2 (CN2), taurine transporter (TauT), PAT1, and phosphorylated Na + / K + / ATPase. The hypotheses are: 1) acute physical exercise increases the uptake of B-alanine by the skeletal muscle; 2) this effect is mediated by the increased activity of the Na + / K + / ATPase pump; 3) this effect, when repeated over five training sessions, results in observable increases in β-alanine → carnosine conversion in skeletal muscle.

DETAILED DESCRIPTION:
B-alanine is a non-essential, non-proteinogenic amino acid found in deficient skeletal muscle concentrations. This deficiency makes B-alanine a rate-limiting factor for carnosine synthesis. B-alanine supplementation is highly efficient in increasing intramuscular carnosine content, leading to improved physical performance, especially in high-intensity exercises (HIIE). It seems that exercise per se can modulate carnosine content; however, it remains uncertain whether physical training or training status can influence B-alanine supplementation responses. Thus, this work aims to assess whether HIIE can increase B-alanine uptake by peripheral tissues and, more specifically, skeletal muscle and increase intramuscular carnosine synthesis. A crossover counterbalanced study will be conducted. The volunteers will be evaluated in two conditions: intake of B-alanine + exercise (B-EX) and B-alanine intake only (B-Ala). The dosage will be 20 mg · kg-1 (powder diluted in water). This process will be divided into two blocks of six days (Thursday to Thursday - without the weekend) with a 4-6 weeks washout. In the B-EX block, a 20-minute HIIE session will be held. Next, B-alanine supplementation will be administered. Immediately after exercise, in a 150-minute rest, collections of venous blood samples will be performed, and the muscle biopsy and urine collection will be collected pre-test and post-test. In the next three days (Thursday to Wednesday), this same protocol will be repeated without blood, muscle, or urine collections. On these days, the B-alanine supplementation will be administrated before and after the protocol (B-EX and B-Ala), in the same dosage of 20mg.kg-1. On the 6th day (Thursday), the complete protocol will be carried out, including the collection of biological materials. In the B-Ala block, the same procedures will be adopted for the B-EX block, with the replacement of the HIIE for 20 minutes of rest sitting on the cycle ergometer. The nutritional parameters will be evaluated during the two blocks by dietary diaries in software (Dietbox) that includes images and the description of all the volunteer food in the day. It will be determined that during the blocks (B-EX and B-ala), the Beta-alanine intake by food is limited to 300mg per day. The analysis of the determination of muscle B-alanine, plasma, and urine, muscle carnosine will be performed by HPLC-ESI + -MS / MS. The gene expression of carnosine-related enzymes and transporters will be analyzed using the real-time PCR technique. The enzymes CARNS1, CN2, TauT, PAT1, and phosphorylated Na + / K + / ATPase will be analyzed using the Western Blot technique. Carnosine synthase activity will be carried out by incorporating [3H] B-alanine acid in the corresponding dipeptide. The analysis of paresthesia's presence and intensity will be through a scale adapted from LINGJÆRDE et al., 1987. The statistical analysis will be performed in the RStudio software and SAS software, using the mixed model to compare muscle, plasma, and urinary variables. Condition (B-Ex vs. B-ala) and time of collection (time) will be fixed factors, while the subjects will be random factors. Data sets containing values obtained at only 2 points in time (e.g., area below the plasma B-alanine curve) will be analyzed using Student's t-test for dependent samples if the data distribution is normal. If the data distribution is not normal, we will use the Wilcoxon sign test for pairs. The normality of data distribution will be assessed qualitatively using Q-Q Plot. Four different covariance matrix structures will be tested for each data set. The Schwarz-Bayesian criterion (lowest BIC value) will be used to select the matrix that best fits each data set. Hypothesis-guided contrast analysis of a single degree of freedom will test specific effects within and between conditions. The size of the Cohen effect (D) will be calculated for all variables. Significance will be accepted if p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* omnivorous diet for> 6 months
* practice physical activities for> 2 h · week-1
* stable body mass (variation <2 kg in the last 30 days)

Exclusion Criteria:

* use of food supplements in the last six months containing β-alanine
* diagnosis of chronic diseases or any other condition that prevents them from performing the proposed procedures
* smoking
* current or past use of anabolic steroids or other ergogenic drugs
* Use of medications that may affect the assessments in this study, including insulin, GH, and thyroid hormone

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2021-05-06 (Actual); Primary Completion 2022-12-23 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Muscle Carnosine after B-alanina supplementation | This evaluation will be carried out with the muscle samples collected on the first and the sixth (last) day of the protocol.
  HPLC-ESI+-MS/MS
Change from Baseline Plasma Beta-alanine after B-alanina supplementation | This evaluation will be carried out with the blood samples collected on the first and the sixth (last) day of the protocol
  HPLC-ESI+-MS/MS

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella B Möller, Msc, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, São Paulo, Brazil